CLINICAL TRIAL: NCT03302676
Title: The Use of Chewing Gum for Xerostomia and Hyposalivation After Radiotherapy for Oral and Oropharyngeal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Cancer Society (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Julie Killerup Kaae, M.D., Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-20160053
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Head and Neck Cancer; Radiation Therapy Complication; Xerostomia; Hyposalivation
Keywords: Saliva substitute
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: 2:1 randomization in favor of chewing gum (intervention)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Patients use tasteless and sugar free chewing gum up to 5 times a day for 1 month.
  Daily registrations in a patient dairy.
  Interventions: Dietary Supplement: Chewing gum
- Control (No Intervention): Patients continue with daily routine to relieve oral discomfort. No chewing gum allowed.

INTERVENTIONS:
Dietary Supplement: Chewing gum
  Arms: Intervention

SUMMARY:
This study evaluates the possible benefits of a tasteless and sugar free chewing gum as a salivary stimulant for head and neck cancer patients treated with curative intended radiotherapy.

DETAILED DESCRIPTION:
Radiation-induced xerostomia and hyposalivation are frequent side effects after completed treatment for oral and oropharyngeal cancers. This may induce eating and swallowing difficulties, compromised oral hygiene, pain in the mouth, or speech deficiencies. As a consequence, quality of life is often impaired for this group of patients even after completing treatment.

This study hypothesize that chewing gum can stimulate salivary flow from the residual functional salivary glands and thereby improving the patient's oral well-being.

Primary endpoint:

- To assess whether the difference between the unstimulated and stimulated salivary flow after a one-month period of using chewing gum will result in improved oral well-being.

Secondary endpoint:

* To assess if unstimulated and stimulated salivary flow differs between the two groups of patients
* To evaluate changes in quality of life with EORTC QLQ H&N-35 for patients using chewing gum
* To evaluate differences in quality of life with EORTC QLQ H&N-35 between the two groups of patients.

All patients who have received curative intended treatment for oral or oropharyngeal carcinomas at the Department of Oncology, Odense University Hospital, will be invited to participate in the study. If the eligibility criteria are met the patient will be randomized 2:1 to either the intervention arm with chewing gum or the control arm with standard oral care. The study intends to include 210 patients in total. Of these, 140 patients in the intervention arm and 70 in the control arm. Recruitment to the study was initiated in September 2016 and is expected to be completed in July 2018.

The duration of the study is one month from inclusion and randomization to final follow up. For all included patients, saliva samples are collected (unstimulated and stimulated sialometry) and the EORTC QLQ H&N-35 questionnaire and a xerostomia specific questionnaire are completed. The patients in the control arm are only introduced to chewing gum at the last follow up visit. In the intervention arm, all patients are instructed to use the chewing gum on a daily basis (preferably 5 times a day) and to make notes in a patient diary to document compliance.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed with oral or oropharyngeal carcinoma
* Received curative intended radiation therapy (primary or postoperative), 60-66Gy including concurrent chemotherapy
* Within 6 to 60 months after radiation therapy
* Complains of xerostomia level 1 (according to Danish Head and Neck Cancer group)
* Written informed consent

Exclusion Criteria:

* Poor teeth condition or full set of dentures
* Recurrence of cancer or palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Salivary flow (intervention arm) | 1 month
  Patients in the intervention arm will experience increase in stimulated salivary flow at follow up as compared to unstimulated salivary flow at baseline.

SECONDARY OUTCOMES:
Salivary flow (both groups of patients) | 1 month
  The difference between unstimulated and stimulated salivary flow will be higher for patients in the intervention arm as compared to the difference in salivary flow for patients in the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Julie K Kaae, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaae JK, Stenfeldt L, Hyrup B, Brink C, Eriksen JG. A randomized phase III trial for alleviating radiation-induced xerostomia with chewing gum. Radiother Oncol. 2020 Jan;142:72-78. doi: 10.1016/j.radonc.2019.09.013. Epub 2019 Oct 9. PMID 31606226